CLINICAL TRIAL: NCT03374072
Title: Engaging Siblings of Adults With Autism in Future Planning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Gael Orsmond, Associate Professor, Boston University Charles River Campus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4366E; R34MH111489 (NIH)
Record Dates: First submitted 2017-12-05; First posted 2017-12-15 (Actual); Results first posted 2023-03-07 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-02

CONDITIONS: Autistic Disorder
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Siblings FORWARD (Experimental): Siblings who participate in the Siblings FORWARD program will participate in telehealth sessions with a community provider. The Siblings FORWARD program includes 6-7 sessions, depending upon whether the autistic adult participates. Siblings work with a program facilitator to develop a future plan of action. They learn communication and problem-solving skills, and about adult service systems.
  Interventions: Behavioral: Siblings FORWARD program
- Information Only Condition (Active Comparator): We will create an online learning module for siblings in the control condition. Siblings in the control condition will be provided with access to the same information about resources for autistic adults provided to participants in the Siblings FORWARD program.
  Interventions: Behavioral: Information Only Condition

INTERVENTIONS:
Behavioral: Siblings FORWARD program — Siblings will participate in a program developed by the researchers designed to engage adults with their autistic sibling and other family members to plan for the future. The Siblings FORWARD program will be implemented by community service providers already working with autistic adults. The program will involve a series individual and joint sessions with siblings and autistic adults using Zoom.
  Arms: Siblings FORWARD
Behavioral: Information Only Condition — Siblings will be provided with online information about services for adults with ASD and future planning.
  Arms: Information Only Condition

SUMMARY:
The goal of this pilot study was to develop and obtain preliminary feasibility and effectiveness data of a telehealth program (Siblings FORWARD) to help siblings of autistic adults work with their families to plan for the future. The main questions it aimed to answer were:

* Is the Siblings FORWARD program feasible to implement via telehealth in the community setting?
* Do siblings benefit from participation in the Siblings FORWARD program?

The Siblings FORWARD program involves 6-7 individualized telehealth sessions with a trained community facilitator. Researchers compared participation in the Siblings FORWARD program to an information-only control condition.

DETAILED DESCRIPTION:
The researchers developed a program to facilitate the engagement of adult siblings to work with their families to plan for the future of their autistic sibling. Siblings FORWARD (Focusing on Relationships, Well-being, and Responsibility aheaD) targeted common barriers to sibling involvement in family future planning, including improving family communication around difficult topics, increasing siblings' knowledge of and confidence in accessing autism service systems, and anticipating and proactively problem-solving barriers to future planning. The Siblings FORWARD program was developed in collaboration with community organizations, with input from siblings, autistic adults, and community providers. Siblings FORWARD was implemented in a community setting, with trained program facilitators. A small randomized controlled trial tested participation in Siblings FORWARD compared to information about services only.

ELIGIBILITY:
Inclusion Criteria:

Siblings of adults with autism spectrum disorder (ASD):

* Have one or more adult brother(s) or sister(s) with ASD who are either biologically related and/or were raised in the same family of origin (e.g., adopted, step, or foster siblings)
* Age 18+.
* English or Spanish fluency.

Autistic Adults:

* Have an ASD diagnosis.
* Have an adult sibling
* Age 21+.
* English or Spanish fluency if verbal.

Exclusion Criteria:

Siblings of autistic adults:

-Siblings will be excluded if they have an ASD diagnosis themselves or if they have any disability that would interfere with their ability to engage meaningfully in future planning for the autistic adult.

Autistic adults:

-None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gael Orsmond, PhD, Principal Investigator — Boston University
Locations (1):
- Boston University, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Information Only Condition: We will create an online learning module for siblings in the control condition. Siblings in the control condition will be provided with access to the same information about resources for autistic adults provided to participants in the Siblings FORWARD program.
  Information Only Condition: Siblings will be provided with online information about services for autistic adults and future planning.
Period: 4 Months
Arm/Group | Siblings FORWARD | Information Only Condition
Started | 10 | 9
Completed | 8 | 9
Not Completed | 2 | 0
Period: 7 Months
Arm/Group | Siblings FORWARD | Information Only Condition
Started | 8 | 9
Completed | 8 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Siblings FORWARD | Information Only Condition | Total
Number analyzed (Participants) | 10 | 9 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.32 (4.96) | 26.37 (3.22) | 25.82 (4.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 2 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 9 | 9 | 18
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 9 | 8 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Quality of Sibling Plan of Action [Mean (Standard Deviation); unit: units on a scale] — Investigator developed. Siblings from both conditions submitted a written plan of action at pre- and post-intervention. The investigators used a template on which siblings detailed their short- and long-term goals with respect to planning for the future with their autistic sibling, and their concrete next steps. Blind ratings of the quality of each plan were conducted, according specific criteria that captured the appropriateness and specificity of the plan. Scores range from 0 to 9, with higher scores representing better quality of plan. Population: One participant from each group did not complete the measure at baseline
  units on a scale
    number analyzed (Participants) | 9 | 8 | 17
    (all) | 7.33 (1.50) | 7.75 (1.48) | 7.53 (1.46)
Family Communication [Mean (Standard Deviation); unit: units on a scale] — Adapted from a measure used by Heller and Caldwell (2006). Siblings rated the frequency with which they have had family discussions about planning for the future of regarding their autistic sibling. Adult sibling participants responded to a 1-item measure scored on a 3-point scale (not discussed at all, discussed somewhat, discussed a great deal). Higher scores reflect more frequent communication.
  units on a scale | 2.10 (0.32) | 1.89 (0.78) | 2.00 (0.58)
Future Planning Self-Efficacy [Mean (Standard Deviation); unit: units on a scale] — Adapted version of the Caregiver Self-Efficacy Scale used by Heller and Caldwell (2006). Sibling participants completed 5 items rated on a 4-point scale (strongly disagree to strong agree). Scores range from 5 to 20, with higher scores indicating higher self-efficacy.
  units on a scale | 14.90 (3.03) | 16.11 (2.67) | 15.47 (2.86)
Sibling Barriers to Future Planning [Mean (Standard Deviation); unit: units on a scale] — Adapted from a measure used by Heller and Caldwell (2006). Sibling participants complete a list of barriers to future planning that includes barriers such as: difficulty finding helpful contact persons within the service system, emotional barriers involved with thinking their parents' mortality, or disagreement with a relative with a disability about the future. Scores ranged from 0 to 12 with higher scores indicating more barriers reported.
  units on a scale | 2.60 (2.91) | 4.33 (3.04) | 3.42 (3.02)
Sibling Knowledge of Adult Services [Mean (Standard Deviation); unit: units on a scale] — Adapted from a measure used by Taylor and Seltzer (2011). Sibling participants rated their knowledge of the 15 services received or needed by their autistic sibling. Siblings rated whether or not their autistic sibling currently receives the services, or if they do not know. If they know that their autistic sibling is not receiving a service, they indicated whether or not that service is needed. Scores ranged from 0 to 15 with higher scores indicating more knowledge.
  units on a scale | 12.20 (2.78) | 10.11 (3.98) | 11.21 (3.47)
Sibling Knowledge of Family Future Plan [Mean (Standard Deviation); unit: units on a scale] — Investigator developed. Siblings completed a checklist of their knowledge (yes/no/ don't know) of whether their family has established: (1) a will, (2) a special needs trust, (3), a financial plan; (4) a letter of intent; (5) a long-term residential plan; or (6) determination of future guardianship. Scores range from 0 to 6 with a high score indicating more areas addressed
  units on a scale | 1.70 (1.89) | 2.22 (2.05) | 1.95 (1.93)

OUTCOME MEASURES:

1. Primary Outcome: Quality of Sibling Plan of Action
Description: Investigator developed. Siblings from both conditions submitted a written plan of action at pre- and post-intervention. The investigators used a template on which siblings detailed their short- and long-term goals with respect to planning for the future with their autistic sibling, and their concrete next steps. Blind ratings of the quality of each plan were conducted, according specific criteria that captured the appropriateness and specificity of the plan. Scores range from 0 to 9, with higher scores representing better quality of plan.
Time Frame: 4 months, 7 months
Population: Missing data from one participant in the Siblings FORWARD condition.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Siblings FORWARD | Information Only Condition
Number analyzed (Participants) | 7 | 9
units on a scale
  4 months | 6.00 (2.38) | 5.44 (2.79)
  7 months | 6.43 (1.51) | 6.56 (1.42)

2. Secondary Outcome: Family Communication About Future Planning
Description: Adapted from a measure used by Heller and Caldwell (2006). Siblings rated the frequency with which they have had family discussions about planning for the future of regarding their autistic sibling. Adult sibling participants responded to a 1-item measure scored on a 3-point scale (not discussed at all, discussed somewhat, discussed a great deal). Higher scores reflect more frequent communication.
Time Frame: 4 months, 7 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Siblings FORWARD | Information Only Condition
Number analyzed (Participants) | 8 | 9
units on a scale
  4 months | 2.13 (0.35) | 2.00 (0.71)
  7 months | 2.00 (0.54) | 1.89 (0.78)

3. Secondary Outcome: Future Planning Self-Efficacy
Description: Adapted version of the Caregiver Self-Efficacy Scale used by Heller and Caldwell (2006). Sibling participants completed 5 items rated on a 4-point scale (strongly disagree to strong agree). Scores range from 5 to 20, with higher scores indicating higher self-efficacy.
Time Frame: 4 months, 7 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Siblings FORWARD | Information Only Condition
Number analyzed (Participants) | 8 | 9
units on a scale
  4 months | 12.38 (3.29) | 15.22 (1.56)
  7 months | 14.00 (1.51) | 15.78 (2.22)

4. Secondary Outcome: Sibling Barriers to Future Planning
Description: Adapted from a measure used by Heller and Caldwell (2006). Sibling participants complete a list of barriers to future planning that includes barriers such as: difficulty finding helpful contact persons within the service system, emotional barriers involved with thinking their parents' mortality, or disagreement with a relative with a disability about the future. Scores ranged from 0 to 12 with higher scores indicating more barriers reported.
Time Frame: 4 months, 7 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Siblings FORWARD | Information Only Condition
Number analyzed (Participants) | 8 | 9
units on a scale
  4 months | 3.38 (2.20) | 4.89 (2.62)
  7 months | 2.88 (1.81) | 4.67 (3.08)

5. Secondary Outcome: Sibling Knowledge of Adult Services
Description: Adapted from a measure used by Taylor and Seltzer (2011). Sibling participants rated their knowledge of the services received or needed by their autistic sibling. The investigators used a list of 15 adult services: physical therapy, occupational therapy, speech and language therapy, psychological or psychiatric services, crisis/intervention services, personal care assistance, agency sponsored recreational or social activities, transportation services, income support, vocational services, respite services, and Medicaid. Siblings rated whether or not their autistic sibling currently receives the services, or if they do not know. If they know that their autistic sibling is not receiving a service, they indicated whether or not that service is needed. Scores ranged from 0 to 15 with higher scores indicating more knowledge.
Time Frame: 4 months, 7 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Siblings FORWARD | Information Only Condition
Number analyzed (Participants) | 8 | 9
units on a scale
  4 months | 14.13 (0.99) | 10.33 (3.24)
  7 months | 14.50 (0.76) | 10.67 (2.83)

6. Secondary Outcome: Sibling Knowledge of Family Future Plan
Description: Investigator developed. Siblings completed a checklist of their knowledge (yes/no/ don't know) of whether their family has established: (1) a will, (2) a special needs trust, (3), a financial plan; (4) a letter of intent; (5) a long-term residential plan; or (6) determination of future guardianship. Scores range from 0 to 6 with a high score indicating more areas addressed
Time Frame: 4 months, 7 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Siblings FORWARD | Information Only Condition
Number analyzed (Participants) | 8 | 9
units on a scale
  4 months | 1.63 (2.20) | 2.78 (2.39)
  7 months | 1.75 (1.98) | 2.44 (1.33)

ADVERSE EVENTS:
Time Frame: 7 months
Arm/Group | Siblings FORWARD | Information Only Condition
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/9
Other Adverse Events (participants affected / at risk) | 0/10 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-02-01): https://cdn.clinicaltrials.gov/large-docs/72/NCT03374072/Prot_SAP_000.pdf
  • Informed Consent Form (2020-09-09): https://cdn.clinicaltrials.gov/large-docs/72/NCT03374072/ICF_001.pdf